CLINICAL TRIAL: NCT02122575
Title: Pilot Study to Evaluate the Effect of Fasting on the NLRP3 Inflammasome
Brief Title: Effect of Fasting on the NLRP3 Inflammasome
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140103; 14-H-0103
Record Dates: First submitted 2014-04-23; First posted 2014-04-24 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Cardiovascular Disease; Inflammatory Disease
Keywords: Inflammasome; Fasting; Sirt3
MeSH Terms: conditions — Cardiovascular Diseases; Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Males and females between the ages of 21 and 37

SUMMARY:
Background:

- Restricting calories can help a person reduce risk factors for heart disease. Researchers have found that not eating or drinking anything but water for 24 hours prevents the activation of a component of the immune system, called the inflammasome. The inflammasome is associated with the development of diabetes and heart disease. Researchers want to learn more about the body s response to fasting.

Objective:

- To explore the benefits of calorie restriction on heart health.

Eligibility:

- Healthy adults ages 21 32 with a body mass index between 26 and 29.

Design:

* Participants will be screened with a medical history, physical exam and blood test.
* Participants will not eat or drink after 10 p.m. before their first visit.
* Participants have breakfast at the clinic. The breakfast will be about 500 calories. Then they will not eat or drink (except water) for 24 hours.
* Participants will return to the clinic the next morning. They will have blood drawn. Then they will have breakfast. Blood will be drawn again at 1 hour and 3 hours after the meal.
* Blood and urine tests at the end of the fast and following the meals will be done to confirm that participants have fasted for the full 24-hour period.

DETAILED DESCRIPTION:
A caloric restricted diet has numerous health effects including the reduction in numerous cardiovascular disease risk factors. The cellular programs activated by caloric restriction are similarly turned on in preclinical studies in response to a 24-hour fast. We have found that a beneficial effect of a 24-hour fasting blunts the activation of a component of the immune system, termed the inflammasome, which is associated with the development of diabetes and atherosclerosis. We would like to study the inflammasome in human blood cells to evaluate whether the beneficial immune effects of fasting/caloric restriction are operational in humans. Blood samples to test the immune response will be collected in subjects after a fixed caloric meal and in response to a 24-hour fast (water intake will not be restricted). The objective of this pilot study is to identify if these immune adaptive pathways can be activated in human subjects as a possible readout to test whether this pathway could be investigated as a therapeutic target to blunt/negate the inflammation associated with nutrient-excess associated diseases such as diabetes and/or atherosclerosis.

ELIGIBILITY:
* INCLUSION CRITERIA:

As this is a pilot study, the age-range and BMI range of subjects will be restricted to potentially reduce metabolic variables associated with a wide age- and BMI-range.

* Males and females between the ages of 21 and 37
* BMI between 23.5 and 29

EXCLUSION CRITERIA:

* Subjects with an acute or chronic illness as per history, on laboratory analysis or due to use of medications
* Subjects taking vitamins or supplements or any medications, except oral contraceptives within 4 weeks of participation into this study.
* BMI <23.5 or >29
* Female subjects who are pregnant or lactating
* Subjects who have donated blood or participated in another clinical trial involving blood draws in the last 8 weeks.
* Subjects who use nicotine products

Ages: 21 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: -Males and females between the ages of 21 and 37@@@-BMI between 23.5 and 29
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-04-21 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Determine whether the NLRP3 inflammasome is blunted by a 24 hours fast in PBMC's from normal volunteers. | 24 hours
  The primary outcome will be the change in IL-1 secretion in response to inflammasome stimulation in PBMC s comparing the fasted response to the fed response. As there are two fed responses, we will initially determine whether inflammasome induction differs between the peak post- prandial insulin effect (1 hr) and the peak post-prandial fatty acid levels (3 hr). The higher mean IL-1 levels between the two fed states will be considered the index fed response and will be compared to the fasting levels as the primary outcome. The comparisons will be performed using paired two-tailed Student t-tests. Significance will be tested at the 0.05 alpha level in this pilot study.

SECONDARY OUTCOMES:
Evaluate whether these effects are associated with activation of the Sirt3 and its canonical mitochondrial adaptive programs. | end of study
  4. Determination of Sirt3 levels and downstream programs in the different nutrient states in PBMC cell samples.
Determine whether serum from subjects in fasted state will blunt the inflammasome compared to serum from the fed stat in a human transformed macrophage cell line. | end of study
  Analysis of difference in inflammasome between the different fed states. Analysis of the inflammasome effect of fed versus fasted serum on transformed THP-1 cells.

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Sack, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Osborn O, Olefsky JM. The cellular and signaling networks linking the immune system and metabolism in disease. Nat Med. 2012 Mar 6;18(3):363-74. doi: 10.1038/nm.2627. PMID 22395709
- [Background] Haneklaus M, Gerlic M, Kurowska-Stolarska M, Rainey AA, Pich D, McInnes IB, Hammerschmidt W, O'Neill LA, Masters SL. Cutting edge: miR-223 and EBV miR-BART15 regulate the NLRP3 inflammasome and IL-1beta production. J Immunol. 2012 Oct 15;189(8):3795-9. doi: 10.4049/jimmunol.1200312. Epub 2012 Sep 14. PMID 22984081
- [Background] Fontana L, Meyer TE, Klein S, Holloszy JO. Long-term calorie restriction is highly effective in reducing the risk for atherosclerosis in humans. Proc Natl Acad Sci U S A. 2004 Apr 27;101(17):6659-63. doi: 10.1073/pnas.0308291101. Epub 2004 Apr 19. PMID 15096581
- [Derived] Traba J, Kwarteng-Siaw M, Okoli TC, Li J, Huffstutler RD, Bray A, Waclawiw MA, Han K, Pelletier M, Sauve AA, Siegel RM, Sack MN. Fasting and refeeding differentially regulate NLRP3 inflammasome activation in human subjects. J Clin Invest. 2015 Nov 3;125(12):4592-600. doi: 10.1172/JCI83260. PMID 26529255
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-H-0103.html